CLINICAL TRIAL: NCT05428202
Title: Phase I Study to Assess Safety, Tolerability and Clinical Benefits of Topically Applied GN-037 Cream in Healthy Volunteers and Patients Diagnosed With Psoriasis
Brief Title: Phase I Study of GN-037 Cream for Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: Monitor CRO (Industry)
Responsible Party: Principal Investigator, Zafer SEZER, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MON839.151.5
Record Dates: First submitted 2022-05-20; First posted 2022-06-23 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Psoriasis
Keywords: Psoriasis; Phase 1 Study; Healthy Volunteers; Patients; Investigational Drug
MeSH Terms: conditions — Psoriasis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Identical tubes with no indicative label, identical creams with similiar texture and odor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GN 037 cream (Experimental): Healthy volunteers will receive GN037 cream in 2 to 1 ration
  Application will be done twice daily, to selected area of body on the fore arm:
  Increasing dosages of dosages: Low dose to a 5 cm2 skin area, Medium dose to15 cm2 skin area, High dose to 30 cm2 skin area
  Psoriatic patients will receive GN037 cream Aplication twice daily, to a selected body target lesion High dose 30 cm2
  Interventions: Drug: GN037
- Placebo Cream (Placebo Comparator): Placebo cream will be applied in 2 to 1 ratio twice daily, to selected area of fore arm.
  Low dose to 5 cm2 skin area, Medium dose 15 cm2 skin area, High dose 30 cm2 skin area
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GN037 — GN-037 cream containing urea, salicylic acid, retinoic acid and clobetasol 17-propionate and matching placebo
  Other Names: Active
  Arms: GN 037 cream
Drug: Placebo — Placebo cream containing base without active ingredients
  Other Names: Placebo Cream
  Arms: Placebo Cream

SUMMARY:
In this Phase I study, three different doses (low, medium and high dose, on the basis of surface area applied) of GN-037 cream (12 volunteers in total) and placebo (6 volunteers in total) will be administered to healthy volunteers. In the active dose arm, 4 healthy volunteers will receive GN-037 cream and 2 healthy volunteers will receive placebo. Randomization in each dose arm will be 2:1.

DETAILED DESCRIPTION:
In this single-center, randomized, double-blind, placebo-controlled, and two-stage Phase I study, it was planned to evaluate the safety, tolerability and clinical efficacy of topically applied GN-037 cream in healthy volunteers and patients diagnosed with plaque psoriasis.

In this Phase I study, three different doses (low, medium and high dose, on the basis of surface area applied) of GN-037 cream (12 volunteers in total) and placebo (6 volunteers in total) will be administered to healthy volunteers. In the active dose arm, 4 healthy volunteers will receive GN-037 cream and 2 healthy volunteers will receive placebo. Randomization in each dose arm will be 2:1.

The study will be performed in two stages; healthy volunteers and patients. After consenting procedures, all subjects will be evaluated for their eligibility for the study. An electronic case report form (e-CRF) specially designed for this study will be used to record the data of the screened volunteers. This e-CRF will assign a volunteer number to each volunteer, as well as providing randomization.

During the screening visit (day 0), a swab for the real-time RT-PCR COVID-19 test will be obtained from all subjects before hospitalization who met the study criteria and gave informed voluntary consent, following the physical examination and screening tests, the volunteers will be interned at the clinic for overnight observation. Hospitalization will be carried out for app 24 hours.

In the healthy subject section of the study, GN-037 cream containing urea, salicylic acid, retinoic acid and clobetasol 17-propionate and matching placebo will be applied to 18 healthy volunteers and will be tested as low dose, medium dose and high dose according to the surface area to be applied in the selected target area. A placebo will be administered to a total of 6 healthy volunteers. All applications will be performed by the investigators during the initial application period and subjects will continue applications as instructed.

GN-037 cream and placebo application will be divided into different stages according to the dose groups specified below, and all volunteers will not be applied on the same day. The study will first start with the administration of low dose GN-037 cream and placebo and will continue through increasing the dosage, hence the applied surface area

* Low dose: 6 healthy volunteers in an area of 5 cm2 in the knee and/or elbow area.
* Medium dose: 6 healthy volunteers on an area of 15 cm2 in the knee and/or elbow area.
* High dose: 6 healthy volunteers will be applied a thin film of GN-037 cream or placebo to an area of 30 cm2 in the knee and/or elbow region, twice a day, morning and evening, for 14 days.

Placebo product will resemble the active products in weight, color and texture.

6 healthy volunteers who were admitted to the clinic at the screening visit will be randomized 2:1 to the low-dose GN-037 cream (n=4) or low-dose placebo (n=2) arm on day 1 of the study. Volunteers in the low dose group will be evaluated for safety data on day 10. If these safety results are found to be appropriate, 6 more healthy volunteers will be recruited for medium dose administration and will be randomized in a 2:1 ratio, with 4 volunteers assigned to the GN-037 cream arm and 2 volunteers to the placebo arm. After safety assessment high dose administration will be initiated. High dose group, will be randomized at a ratio of 2:1; as active:placebo and after final safety evaluation patients with plaque psoriasis (n=6) will be included in the study. All inclusion and efficacy/safety evaluations will be performed by a dermatologist.

All subjects will be treated for 14 days (active and placebo) and a final safety evaluation will be performed on day 19. Study drugs will be collected on this visit and the cream usage will be measured by weighing the used cream tubes. On day 28, a telephone visit will be performed for final safety evaluation.

ELIGIBILITY:
Inclusion Criteria: Healthy Volunteers

1. Male and female healthy volunteers aged 18-65 years*
2. Volunteers who were informed about participation in the study and agreed to give their written informed consent.
3. Volunteers with negative qPCR SARS-CoV-2 result in nasopharyngeal or sputum samples
4. Volunteers in good general health (without any known disease in the history and physical examination in the 14 days before participating in the study)
5. Volunteers with negative HIV, Hepatitis B and C tests
6. Volunteers with negative alcohol breath test
7. Volunteers with negative urine addictive drug screening test (amphetamine, barbiturate, benzodiazepine, cannabinoid, cocaine, opiate)
8. Volunteers who agreed not to be exposed to the direct sun light during the study
9. Female volunteers of childbearing potential must have a negative pregnancy test at the screening visit and must agree to use an effective method of contraception throughout the study
10. Volunteers who can comply with all scheduled visits, laboratory tests and other study procedures * The principal investigator will take the necessary measures to ensure that the representation

Exclusion Criteria Healthy Volunteers

1. Subjects with known hypersensitivity to any component of the study drug
2. Female volunteers who are pregnant or breastfeeding or have a positive pregnancy test
3. Volunteers with a history of chronic or acute infections requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks prior to the screening visit
4. Patients with skin atrophy, pigmentation or extensive scarring that would preclude study evaluation at targeted treatment sites
5. Patients with other inflammatory skin disease (eg, atopic dermatitis, contact dermatitis, eczema, tinea corporis) that, in the investigator's opinion, may affect study evaluations at targeted treatment sites
6. Volunteers using moisturizing or skin softening ointment/lotion/cream on their intended treatment site within 3 days prior to enrollment in the study.
7. Volunteers who cannot come to the study center for follow-up visits
8. Volunteers taking part in another clinical study concurrently
9. Volunteers with positive urine addictive drug screening test and/or alcohol test

Inclusion Criteria For psoriatic patients

1. Male and female patients aged 18-65 years*
2. Patients who were informed about participation in the study and agreed to give their written informed consent.
3. Patients with negative qPCR SARS-CoV-2 result in nasopharynx or sputum samples
4. Patients diagnosed with plaque psoriasis by a dermatologist at least 6 months before inclusion in the study
5. Patients whose lesions are less than 5% of the body surface area (BSA)
6. Patients who did not receive local or systemic treatment for plaque psoriasis, or who received the last psoriasis treatment 28 days or more before
7. Patients who are confirmed to be healthy by medical history and physical examination and who do not have any clinically significant disease/condition other than plaque psoriasis that could affect the study evaluation.
8. Patients with disease severity with Physician's Global Assessment (IGA) score ≥3 (moderate) as an overall assessment of all lesions to be treated
9. Patients with negative HIV, Hepatitis B and C tests
10. Patients with negative alcohol breath test
11. Patients with negative urine addictive drug screening test (amphetamine, barbiturate, benzodiazepine, cannabinoid, cocaine, opiate)
12. Patients who agreed not to be exposed to the sun during the study
13. Female patients of childbearing potential must have a negative pregnancy test at the screening visit and must agree to use an effective method of contraception throughout the study
14. Patients who can comply with all scheduled visits, laboratory tests, and other study procedures * The principal investigator will take the necessary measures to ensure that the representation of females and males is equal.

Exclusion criteria For psoriatic patients

1. Patients with known hypersensitivity to any component of the study drug
2. Pregnant or lactating or female patients with a positive pregnancy test
3. Patients who require any other medication (topical or systemic) that may affect the course of the disease during the study period (eg antibiotics, antihistamines)
4. Patients with a history of chronic or acute infections requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks prior to the screening visit
5. Patients with skin atrophy, pigmentation, or extensive scarring that would preclude evaluation of study drug efficacy at targeted treatment sites
6. Patients with other inflammatory skin disease (eg, atopic dermatitis, contact dermatitis, eczema, tinea corporis) that, in the investigator's opinion, may affect study evaluations at targeted treatment sites
7. Patients diagnosed with pustular, guttate, inverse, exfoliative or erythrodermic psoriasis at targeted treatment sites
8. Patients with a history of psoriasis unresponsive to topical treatments
9. Patients who used moisturizer or skin softening ointment/lotion/cream to the intended treatment areas within 3 days prior to enrolling in the study.
10. Patients who cannot come to the study center for follow-up visits
11. Patients taking part in another clinical study concurrently
12. Patients with positive urine addictive drug screening test and/or alcohol test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Severity of Adverse Events and Serious Adverse Events. | 28 days
  Severity of all Adverse Events (AEs) and Serious Adverse Events (SAEs) that occur during the whole trial including the observational period (AEs and SAEs include but not limited to comorbidities, such as hypertension, diabetes, and cardiovascular diseases).

SECONDARY OUTCOMES:
Percent Change From Baseline in Total Plaque Severity Score in Psoriasis Patients From baseline at days 6 and 14 with GN-037 cream application. | 19 days
  Difference in least squares mean percent change from baseline at days 6 and 14 in total plaque severity score (TPSS) with GN-037 cream application. For TPSS, all target lesions were scored individually for signs of induration, scaling, and erythema using a 5-point severity scale: 0 = none; 1 = mild; 2 = moderate; 3 = severe; 4 = very severe. A negative percent change indicates better outcome.
Percent Change From Baseline in Target Plaque Area in Psoriasis Patients From baseline at days 6 and 14 with GN-037 cream application. [ Time Frame: 19 days ] | 19 days
  Difference in least squares mean percent change from baseline at days 6 and 14 in target plaque area (TPA) with GN-037 cream application. Target plaque area (cm2) was determined by multiplying the longest diameter (cm) of the target plaque by the widest perpendicular diameter (cm) (perpendicular to the longest diameter of the target plaque). A negative percent change indicates mild disease
Difference in Psoriasis Area Severity Index (PASI) From baseline at days 6 and 14 with GN-037 cream application. | 19 days
  The PASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema (redness), induration (plaque thickness), and scale, and the extent of %Body Surface Area (BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0 to 4) and the %BSA affected is scored on a 7-point scale (0 to 6) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease. PASI is a static assessment made without reference to previous scores.
Change in Physician Global Assessment (PGA) score From Baseline achieved at days 6 and 14 with GN-037 cream application. | 19 days
  The PGA is a clinical tool for assessing the current state/severity of a participant's psoriasis at a given timepoint. It is a static 6-point (0-5) morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, scaling, and plaque thickness/elevation as guidelines. Higher PGA scores represent more severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: Oğuz Akbaş, MD, Study Director — Monitor CRO
Locations (1):
- Erciyes University IKUM Center, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sezer Z, Inal A, Cinar SL, Mazicioglu MM, Altug S, Karasulu HY, Diril M, Mehmetoglu Al A, Kozlu S, Ulu N. Safety and Efficacy of a Novel Combination Cream (GN-037) in Healthy Volunteers and Patients with Plaque Psoriasis: A Phase 1 Trial. Dermatol Ther (Heidelb). 2023 Jul;13(7):1489-1501. doi: 10.1007/s13555-023-00939-7. Epub 2023 Jun 10. PMID 37300792